CLINICAL TRIAL: NCT00174629
Title: Open-Label, Cooperative, Randomized, Multicenter Phase III Study on the Use of Cisplatin Resistant Genotype (ERCC1 Over-Expression) in Tumor RNA to Customize Chemotherapy in Stage IV-IIIB (Malignant Pleural Effusion) Non-Small-Cell Lung Cancer Patients
Brief Title: GILT Docetaxel - Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAX_ES1_302
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Gemcitabine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: docetaxel/gemcitabine
- 2 (Active Comparator)
  Interventions: Drug: Docetaxel/DDP

INTERVENTIONS:
Drug: Docetaxel/DDP
  Arms: 2
Drug: docetaxel/gemcitabine
  Arms: 1

SUMMARY:
Primary Objective:

* To compare response rate between genotypic groups and control group.

Secondary Objective:

* To determine the safety, time to treatment failure and survival in control and genotypic arms.

ELIGIBILITY:
Inclusion Criteria:

Patients must be/have:

* histologically confirmed non-small cell lung cancer (squamous cell carcinoma, large cells or adenocarcinoma; it is recommended to provide the full paraffin-embedded block or at least 5 5 sections obtained from the primary tumor, recurrence or metastasis, not stained, fixed in formalin/embedded in paraffin, mounted on slides (10 micron sections), as well as two serum samples in two 10-ml tubes and two blood samples (see appendix X);
* unresectable metastatic (stage IV or IIIB malignant pleural effusion) NSCLC;
* WHO performance status < 2;
* Adequate bone marrow, hepatic and renal functions, assessed during the previous 14 days, that should be shown by the following characteristics:

  * hemoglobin > or = 10g/dl and no blood cell transfusion within the previous 2 weeks;
  * absolute neutrophil count > 2.0 10^9 cells/l;
  * platelet count > or = 100.10^9 cells/l;
  * no evidence of myelodysplastic syndrome or abnormal bone marrow reserve;
  * creatinine < or = 1.5 x UNL or creatinine clearance > or = 60 ml/min (real or calculated);
  * total bilirubin < or = UNL;
  * ASAT (SGOT) and/or ALAT (SGPT) < or = 1.5 x UNL;
  * alkaline phosphatases < or = 5 x UNL;
  * serum calcium < or = 1.1 x UNL;
* at least one measurable lesion;
* previous surgery intervention (more than 30 days before inclusion in the study) is allowed but metastatic disease must be demonstrated;
* previous radiotherapy is allowed if:

  * less or equal to 10% of bone marrow has been irradiated
  * end of radiotherapy 21 days or more prior to inclusion in the study;
  * patient has fully recovered from all toxic effects;
  * at least one of the measurable target lesions for evaluation of tumor response has not been irradiated;
* the patient must be accessible for treatment and follow-up. The patient entered into this trial must be treated and followed up at the participating center;
* life expectancy > or = 12 weeks;
* The initial diagnostic procedures should be performed during the 4 weeks prior to the randomization.

Exclusion Criteria:

* pregnant or lactating women (women of childbearing potential must use adequate contraception);
* prior systemic chemotherapy or immunotherapy for NSCLC, even as neoadjuvant or adjuvant therapy;
* prior malignancies, except cured non-melanoma skin cancer, curatively treated in situ carcinoma of the cervix or other cancer curatively treated and with non-evidence of disease for at least 5 years;
* history or clinical symptomatic brain or leptomeningeal metastases;
* current peripheral neuropathy and neurohearing > or = NCIC-CTG grade 2 except if due to trauma;
* other serious illness or medical condition, including:

  * congestive heart disease; prior myocardial infarction within 6 months;
  * history of significant neurologic or psychiatric disorders that would inhibit their understanding and giving of informed consent;
  * infection requiring I.V. antibiotics and tuberculosis under treatment ongoing at study entry;
  * untreated superior vena cava syndrome;
  * active peptic ulcer; unstable diabetes mellitus or other contraindication to high dose corticotherapy such as herpes, herpes zoster, cirrhosis;
* hypercalcemia requiring therapy;
* preexisting ascitis and/or clinical significant pericardial effusion;
* patients whose lesion(s) are assessable only by radionuclide scan;
* history of allergy to drugs containing the excipient TWEEN 80®;
* concurrent treatment with other investigational drugs;
* participation in a clinical trial of one or more investigational agents (i.e. antibiotic) or devices within 30 days of study entry.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2001-06; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete plus partial responses) between the genotypic group and the control group using an intent-to-treat analysis.

SECONDARY OUTCOMES:
Time to treatment failure and survival | calculated from the registration date until progression or death, respectively
Clinical and laboratory toxicities graded according to NCIC-CTG Expanded Common Toxicity Criteria. | before each cycle
Adverse events not reported in NCIC-CTG Expanded Common Toxicity Criteria will be graded as mild, moderate, severe, and life threatening. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Aussel, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Geneva, Switzerland